CLINICAL TRIAL: NCT06500442
Title: A Phase 1 Study of NEU-111 Administered Orally to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Healthy Volunteers
Brief Title: A Study to Assess NEU-111 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuron23 Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-111-UC101
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEU-111 (Experimental): Part A: Single-ascending dose cohorts; Part B: Multiple-ascending dose cohort (10 days)
  Interventions: Drug: NEU-111
- Placebo (Placebo Comparator): Part A: Single-ascending dose cohorts; Part B: Multiple-ascending dose cohorts (10 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NEU-111 — Oral Doses
  Arms: NEU-111
Drug: Placebo — Oral Doses
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose (SAD), multiple ascending dose (MAD), of orally administered NEU-111 in healthy subjects.

DETAILED DESCRIPTION:
Up to five (5) single-ascending oral doses will be administered to 40 healthy adult male or female subjects, (aged 18-64 years, inclusive). Escalation to the next higher dose level may occur only after evaluation of the safety and available PK results of the previous dose level (at least 6 evaluable subjects). Within each cohort, 6 subjects will receive one dose of NEU-111, and 2 subjects will receive one dose of matching placebo. Dose levels may be revised based upon available safety and PK data.

Multiple ascending oral doses will be administered up to 24 healthy subjects, (aged 18-64 years, inclusive) in 3 sequential dosing groups (8 subjects in each dosing group). Six (6) subjects will receive NEU-111 and two (2) subjects will receive matching placebo in each dosing group (cohort) for 10 days. Escalation to the next higher dose level may occur only after evaluation of the safety and PK results of the previous dose level (at least 6 evaluable subjects). Dose levels may be revised based upon available safety and PK data.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

Subjects for standard cohorts must be 18-64 years, inclusive, at the time of signing the informed consent; Subjects who are in good general health with no clinically relevant abnormalities based on the medical history, physical examinations, neurological examinations, clinical laboratory evaluations (hematology and clinical chemistry) Subjects who have a body mass index (BMI) of 18-32 kg/m2(inclusive);

Male subjects are eligible to participate if they are rendered surgically sterile (at least 6 months), or agree to the following during the study and for at least 30 days after the last dose of study drug:

• Refrain from donating sperm;

AND, either:

Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; OR Agree to use a male condom (contraception/barrier) and should also be advised of the benefit for a female partner to use an acceptable, highly effective method of contraception as a condom may break or leak when having sexual intercourse;

Female subjects are eligible to participate if they are not pregnant or breastfeeding, subject to one of the following:

Women of childbearing potential (WOCBP), defined as women physiologically capable of becoming pregnant, must have a negative serum pregnancy test at the Screening visit and a negative urine pregnancy test on Day -1; WOCBP must agree to use an acceptable, highly effective contraceptive method from Screening until 30 days after the last dose of study treatment (see Section 11.3); OR Menopausal women must have an elevated serum follicle-stimulating hormone level (FSH) level at Screening; if the FSH is not elevated, they are considered to be of childbearing potential (unless permanently sterile) and must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1;

Exclusion Criteria:

History of clinically significant hematological, renal, pancreatic, gastrointestinal, hepatic, cardiovascular, metabolic, endocrine, immunological, allergic disease, or other major disorders Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia; Use of or plans to use systemic immunosuppressive (e.g., corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 3 months prior to the first study drug administration;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of single and multiple oral doses of NEU-111 in healthy subjects | Up to 10 days of dosing
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
PK Parameter | Up to 10 days of dosing
  The maximum concentration (Cmax) at steady state in plasma
PK Parameter | Up to 10 days of dosing
  The area under the concentration-time curve from zero to infinity (AUC0-inf) in plasma
PK Parameter | Up to 10 days of dosing
  The time to reach maximum concentration (tmax) in plasma
PK Parameter | Up to 10 days of dosing
  Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) in plasma
PK Parameter | Up to 10 days of dosing
  Apparent terminal elimination half-life (t1/2) in plasma
PK Parameter | Up to 10 days of dosing
  The terminal elimination rate constant (λZ) with the respective half-life (t½) in plasma
PK Parameter | Up to 10 days of dosing
  The oral clearance (CL/F)
PK Parameter | Up to 10 days of dosing
  The volume of distribution (Vd/F)
PK Parameter | Up to 10 days of dosing
  The area under the concentration-time curve over a dosing interval (AUC0-τ) in plasma (multiple dosing only)

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided